CLINICAL TRIAL: NCT02849691
Title: Plasma Dipeptidyl-peptidase-4 Activities With No-reflow and Bleeding
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Jing Wei, Dr., Chinese PLA General Hospital
Other Study IDs: DPP4a-noreflow
Record Dates: First submitted 2016-07-24; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Dipeptidyl-peptidase-4; STEMI; PCI; No-reflow; Bleeding
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Quartile 1: Quartile 1 of plasma DPP4 activity
- Quartile 2: Quartile 2 of plasma DPP4 activity
- Quartile 3: Quartile 3 of plasma DPP4 activity
- Quartile 4: Quartile 4 of plasma DPP4 activity

SUMMARY:
Dipeptidyl-peptidase-4 (DPP4) is an important regulator of incretins and inflammation, and participates in the pathophysiological process of acute myocardial infarction (AMI). However clinical data of DPP4a in AMI patients is sparse. This study was to investigate the role of plasma DPP4 activity (DPP4a) in patients with ST-segment elevation myocardial infarction (STEMI) treated with percutaneous coronary intervention (PCI). This was a analysis of consecutive patients conducted at a tertiary referral center from January 2014 to October 2015. The investigators included 747 STEMI-patients, treated with PCI from January 2013 to October 2015. Blood samples were collected immediately at admission. The patients were divided into four groups according to DPP4a quartile.

DETAILED DESCRIPTION:
ST-segment elevation myocardial infarction (STEMI) is an acute manifestation of coronary heart disease, remaining a frequent cause of death.A better understanding of risk factors and pathogenic mechanisms underlying STEMI may help improve the prognosis and life quality of these patients.Dipeptidyl peptidase 4 (DPP4) is an exopeptidase expressed on the surface of diverse cells, cleaving off amino-terminal dipeptides with either L-proline, L-alanine or serine at the penultimate position. As a cell surface protein, it participates in immune regulation, signal transduction and apoptosis. DPP4 also circulates as a soluble form in the plasma. Soluble DPP4 came from either membrane type clearance or secreted by cells like endothelial cells, with enzymatic activity. Plasma DPP4 activity (DPP4a) are elevated in several diseases, including type 2 diabetes, obesity, atherosclerosis and osteoporosis. Basic studies have showed that DPP4 inhibition leads improved survival and heart function after cardiac ischemia-reperfusion (I/R) injury, and this is partly due to activation of AKT (pAKT), pGSK3 and ANP pathways. Also inhibition of DPP4 can alleviate atherosclerosis and heart failure. Accordingly, one could hypothesize that high DPP4a may worsen myocardial I/R injury, causing poorer cardiovascular outcomes. However, no study has evaluated whether DPP4a is associated with adverse clinical outcomes in STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of STEMI and needed PCI

Exclusion Criteria:

* patients with cancer
* patients who used DPP4 inhibitor
* patients who used GLP1 analogue

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PLA general hospital (PLAGH) is a large national tertiary-care center in the Beijing, China. The investigators enrolled all patients consecutively hospitalized in PLAGH, with a diagnosis of STEMI and needed PCI.
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
a change in the prevalence of no-reflow | immediately after PCI
  TIMI flow grade of <3 with a myocardial blush grade of 0-1 was defined as angiographic no-reflow

SECONDARY OUTCOMES:
in-hospital major adverse cardiac or cerebrovascular events | up to 2 week after PCI (until discharge)
  the composite of death, nonfatal MI, or stroke
in-hospital complications | up to 2 week after PCI (until discharge)
  defined as acute heart failure, atrial fibrillation, chest pain or re-acute myocardial infarction, complete atrioventricular block, cerebrovascular disease, ventricular fibrillation or ventricular tachycardia
in-hospital major bleeding | up to 2 week after PCI (until discharge)
  defined as absolute hemoglobin drop (baseline to nadir)≥4g/dl, intracranial hemorrhage, retroperitoneal hemorrhage, use of red blood cell transfusion in patients with a baseline hemoglobin ≥9.0 g/dl, and use of red blood cell transfusion among patients with a baseline hemoglobin <9.0 g/dl and a witnessed bleeding event

REFERENCES:
- [Background] Windecker S, Bax JJ, Myat A, Stone GW, Marber MS. Future treatment strategies in ST-segment elevation myocardial infarction. Lancet. 2013 Aug 17;382(9892):644-57. doi: 10.1016/S0140-6736(13)61452-X. PMID 23953388
- [Background] Zhong J, Rajagopalan S. Dipeptidyl Peptidase-4 Regulation of SDF-1/CXCR4 Axis: Implications for Cardiovascular Disease. Front Immunol. 2015 Sep 25;6:477. doi: 10.3389/fimmu.2015.00477. eCollection 2015. PMID 26441982
- [Background] Zhong J, Maiseyeu A, Davis SN, Rajagopalan S. DPP4 in cardiometabolic disease: recent insights from the laboratory and clinical trials of DPP4 inhibition. Circ Res. 2015 Apr 10;116(8):1491-504. doi: 10.1161/CIRCRESAHA.116.305665. PMID 25858071
- [Background] Connelly KA, Zhang Y, Advani A, Advani SL, Thai K, Yuen DA, Gilbert RE. DPP-4 inhibition attenuates cardiac dysfunction and adverse remodeling following myocardial infarction in rats with experimental diabetes. Cardiovasc Ther. 2013 Oct;31(5):259-67. doi: 10.1111/1755-5922.12005. PMID 22963483
- [Background] Shigeta T, Aoyama M, Bando YK, Monji A, Mitsui T, Takatsu M, Cheng XW, Okumura T, Hirashiki A, Nagata K, Murohara T. Dipeptidyl peptidase-4 modulates left ventricular dysfunction in chronic heart failure via angiogenesis-dependent and -independent actions. Circulation. 2012 Oct 9;126(15):1838-51. doi: 10.1161/CIRCULATIONAHA.112.096479. Epub 2012 Oct 3. PMID 23035207